CLINICAL TRIAL: NCT02385851
Title: A Randomized, Double-Blind, Crossover Study to Compare the Pharmacokinetic and Pharmacodynamic Biosimilarity of CHS-1701 (Coherus Pegfilgrastim) With Neulasta® in Healthy Subjects
Brief Title: Comparison of the Pharmacokinetic and Pharmacodynamic Biosimilarity of CHS-1701 (Coherus Pegfilgrastim) With Neulasta® (Pegfilgrastim)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: CHS-1701-03
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Bioequivalence
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHS-1701/Neulasta (Experimental): CHS-1701 followed by Neulasta (crossover)
  Interventions: Drug: CHS-1701; Drug: Pegfilgrastim
- Neulasta/CHS-1701 (Experimental): Neulasta followed by CHS-1701 (crossover)
  Interventions: Drug: CHS-1701; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: CHS-1701
Drug: Pegfilgrastim
  Other Names: Neulasta

SUMMARY:
This is a randomized, double-blind, single-dose, 2-period crossover study in healthy subjects to assess PK, PD, and safety (including immunogenicity) of a single 6 mg subcutaneous (SC) injection of CHS-1701 compared with a single 6 mg SC dose of Neulasta®.

DETAILED DESCRIPTION:
This is a randomized, double-blind, single-dose, 2-period crossover study in healthy subjects to assess PK, PD, and safety (including immunogenicity) of a single 6 mg subcutaneous (SC) injection of CHS-1701 compared with a single 6 mg SC dose of Neulasta®.

After screening, eligible subjects will be randomly assigned to 1 of 2 treatment sequences; CHS-1701 followed by Neulasta® (Sequence A) or Neulasta® followed by CHS-1701, Sequence B). Treatments will be spaced by a minimum of 6 weeks apart (but no more than 8 weeks). Subjects will be admitted to the Clinical Pharmacology Unit (CPU) on Day -1 (Period 1) and will be confined through Hour 96 postdose (a total of approximately 4.5 days and 5 nights). Blood samples will be collected at specified time points postdose for plasma PK and PD measurements and the subjects will be closely monitored for safety. Following discharge on the morning of Day 5 (Period 1) subjects will return to the clinic for additional PK, PD and safety follow up--daily through Day 9 and at stated interval time points thereafter.

The single dose of the alternate blinded study drug will be given after 6 (but no more than 8) weeks of observation and washout and the above procedures will be repeated (Period 2). A Follow up Visit will take place 41 (±1) days after the second dose.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female of ages 18 to 50 inclusive
2. Body weight > 50 kg (110 lb.) and body mass index between 18 and 32 kg/m2 inclusive
3. Medically healthy with clinically insignificant findings based on medical history, 12-lead ECG, and physical examination
4. Negative urine pregnancy test in women of childbearing potential

Exclusion Criteria:

1. Previous exposure to pegfilgrastim or filgrastim, or known allergy to PEG (polyethylene glycol)
2. Chemistry and hematology values outside protocol specified range
3. Current or previous cancer, diabetes, or any clinically significant cardiovascular, metabolic, renal, hepatic, gastrointestinal, hematologic, respiratory, dermatological, neurological, psychiatric, or other disorder
4. History of chronic or acute respiratory illness within the past 4 weeks
5. Positive urine drug or alcohol screen or unwillingness to abstain from alcohol or recreational drugs for the duration of study participation
6. No prescription or nonprescription drugs during the study
7. Participation in an investigational clinical study within 30 days prior to screening
8. Known or suspected allergic reaction to latex

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Biosimilarity as measured by absolute neutrophil count (ANC) | 84 Days
  The primary objective of this study is to assess the biosimilarity of CHS-1701 with Neulasta® based on the pharmacokinetics (PK) of pegfilgrastim and the pharmacodynamic (PD) response as measured by absolute neutrophil count (ANC).

SECONDARY OUTCOMES:
PK Profile: Cmax (tmax), AUC0-t, and t1/2 | 84 Days
  Characterization of the PK profile of CHS-1701 using standard parameters (Cmax (tmax), AUC0-t, and t1/2)
Safety Profile as assessed by clinical adverse events (AEs), laboratory variables, vital signs, incidence of antidrug antibodies (ADAs), and local injection site reactions (ISRs). | 84 Days
  Characterization of the safety profile and tolerance of CHS-1701, as assessed by clinical adverse events (AEs), laboratory variables, vital signs, incidence of antidrug antibodies (ADAs), and local injection site reactions (ISRs).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Finck, MD, Study Director — Coherus Oncology, Inc.
Locations (1):
- ICON, San Antonio, Texas, United States

REFERENCES:
- [Derived] Civoli F, Finck B, Tang H, Hodge J, O'Kelly H, Vexler V. Biosimilar Pegfilgrastim-cbqv Demonstrated Similar Immunogenicity to Pegfilgrastim in Healthy Subjects Across Three Randomized Clinical Studies. Adv Ther. 2022 Mar;39(3):1230-1246. doi: 10.1007/s12325-021-02024-x. Epub 2022 Jan 16. PMID 35034311